CLINICAL TRIAL: NCT05968729
Title: Assessment of Gait Adaptation Due to an Asymmetric Walking Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kristin Morgan, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H21-0176; K01AR079043 (NIH)
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.25 m/s asymmetric session first (Active Comparator): Participants will perform three 15-minute sessions of walking with a 0.25 m/s asymmetric walking gait speed difference where one limb is set at 1.0 m/s and the other limb is set at 1.25 m/s. Each of these sessions will be followed by 5-minute de-adaptation sessions where they will perform a symmetric walking trial at 1.0 m/s.
  Interventions: Other: Active Comparator: 0.25 m/s asymmetric session first
- 0.50 m/s asymmetric walking session first (Active Comparator): Participants will perform three 15-minute sessions of walking with a 0.50 m/s asymmetric walking gait speed difference where one limb is set at 1.0 m/s and the other limb is set at 1.5 m/s. Each of these sessions will be followed by 5-minute de-adaptation sessions where they will perform a symmetric walking trial at 1.0 m/s.
  Interventions: Other: Active Comparator: 0.50 m/s asymmetric session first

INTERVENTIONS:
Other: Active Comparator: 0.25 m/s asymmetric session first — Participants will first perform an asymmetric walking trial where the between-limb gait speed difference is 0.25 m/s on day one. On the second day, participants will perform an asymmetric walking trial where the between-limb gait speed difference is 0.50 m/s.
  Arms: 0.25 m/s asymmetric session first
Other: Active Comparator: 0.50 m/s asymmetric session first — Participants will first perform an asymmetric walking trial where the between-limb gait speed difference is 0.50 m/s on day one. On the second day, participants will perform an asymmetric walking trial where the between-limb gait speed difference is 0.25 m/s.
  Arms: 0.50 m/s asymmetric walking session first

SUMMARY:
The purpose of this work is to conduct a comparative research-focused study to evaluate the effectiveness of how purposefully induced asymmetric walking protocols restore healthy, symmetric limb loading in individuals following post-anterior cruciate ligament reconstruction (ACLR) surgery. Additionally, computational modeling and machine learning to model knee loading in the clinic to determine the optimal asymmetric walking protocol to restore healthy gait in post-ACLR individuals.

DETAILED DESCRIPTION:
This is an intervention study in which participants will be randomized as to the order in which each of the two sessions are completed. Forty post-ACLR will who present with between-limb gait differences will perform two asymmetric walking sessions where they will walk with between-limb gait speed differences of 0.25 m/s and 0.50 m/s at three 15-minute intervals to evaluate the restoration of healthy gait. Post-ACLR participants will perform an asymmetric walking intervention protocol session on two different days. On one day they will perform the protocol with a 0.25 m/s between-limb difference and on a separate day they will perform the protocol with a 0.50 m/s between limb difference. For the 0.25 m/s condition, one limb will be set to 1.0 m/s and the other 1.25 m/s (i.e., 1.0 m/s - 1.25 m/s). Similarly, for the 0.50 m/s condition, one limb will be set to 1.0 m/s and the other 1.50 m/s (i.e., 1.0 m/s - 1.50 m/s). Each participant will perform both the 0.25 m/s and 0.50 m/s protocols on separate days, and we will randomize who performs which protocol first or second. At least 3 weeks must pass between the two one-day sessions. Patient-specific simulations will be generated in OpenSim for each of the 40 post-ACLR individuals to assess differences in knee joint loading. Together with machine learning, these models will help evaluate the effectiveness of the asymmetric walking protocol in reducing detrimental knee loading. The study team hypothesizes that the 0.50 m/s perturbation will produce a larger reduction in between-limb asymmetry than the 0.25 m/s perturbation and reduce detrimental knee loading.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and speak English
2. Age 18 - 30 years old
3. Undergone ACLR surgery at the UConn Musculoskeletal Institute
4. Must not have any concomitant surgeries or injuries
5. Must be cleared to return-to-sport by a physician after they have completed rehabilitation
6. Must be within 1 month of having been cleared for return-to-sport
7. Must present with between-limb gait differences in load rate greater than 10%

Exclusion Criteria:

1. Participants who have any recent inflammation, bleeding disorders, active bleeding, or infection within the lower limbs.
2. History of injuries to their patellar tendon
3. Cannot walk for extended periods of time
4. Cannot have had any back and/or lower extremity injury that affects their ability to move.
5. Cannot have difficulty or pain with walking, raising your arms, jogging, or jumping
6. Must not be allergic to tape.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Loading Rate | Screening, Baseline, and Post-Treatment (immediately following the completion of the second session)
  The rate at which the force is generated (Body Weight/sec). A decrease in loading rate would suggest that the participants adopted improved motor control while an increase would reflect impaired of motor control.
Change in Peak Vertical Ground Reaction Force | Baseline, Post-Treatment (immediately following the completion of the second session)
  The largest force (newtons) produced during stance. An increase in force would that the participants are not properly engaging their muscles to control their movement.
Change in Stride Time | Baseline, Post-Treatment (immediately following the completion of the second session)
  The time (seconds) measure from initial contact on the foot to the next initial contact on the same foot. A reduction in stride time would indicate that the participants are walking faster and more comfortable applying force to their limb during walking. An increase in walking speed, suggests that the participants are uncomfortable applying force to their limb.
Change in Knee Loading | Baseline, Post-Treatment (immediately following the completion of the second session)
  The forces (newtons) experienced at the knee. An increase in knee loading would indicate that they participants are unable to properly support their knee during walking, while a reduction in knee loads would indicate the participants are engaging the appropriate muscles to support their knee during walking.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Morgan, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No